CLINICAL TRIAL: NCT03486275
Title: Development and Evaluation of Hygie, a New Serious Game for Continuing Medical Education of General Practitioners: a Randomized Trial
Brief Title: Development and Evaluation of Hygie, a New Serious Game for Continuing Medical Education of General Practitioners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hygie (Other)
Responsible Party: Principal Investigator, Louis-Baptiste Jaunay, Researcher, Hygie
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Hygie1
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: CONTINUING MEDICAL EDUCATION
Keywords: GENERAL PRACTICE; SERIOUS GAME; EVIDENCE BASED MEDICINE; RANDOMIZED CONTROLLED TRIAL; PEDAGOGY

STUDY DESIGN:
Intervention Model Description: randomized trial comparing the learning provided by a week of access to the game Hygie or source articles
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded randomized trial : Participants do not know their assignment group. The questionnaires, identical in both groups, were completed by the participants and blinded from their assignment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hygie game (Active Comparator): Prototype video game called Hygie on the 5 most common reasons of consultation in general practice using 9 articles from independent journals based on evidence (reviews by Prescrire and Minerva).
  Interventions: Device: Hygie
- Source articles (Active Comparator): 9 articles from independent journals based on evidence (reviews by Prescrire and Minerva)
  Interventions: Device: Source articles

INTERVENTIONS:
Device: Hygie — Prototype video game called Hygie, accessible on the Internet, on the 5 most common reasons of consultation in general practice using 9 articles from independent journals based on evidence (reviews by Prescrire and Minerva).
  Arms: Hygie game
Device: Source articles — 9 articles from independent journals based on evidence (reviews by Prescrire and Minerva), about the 5 most common reasons of consultation in general practice, accessible on the Internet.
  Arms: Source articles

SUMMARY:
We produced a prototype video game called Hygie on the 5 most common reasons of consultation in general practice using 9 articles from independent journals based on evidence (reviews by Prescrire and Minerva). We then carried out a randomized trial comparing the learning provided by a week of access to the game versus source articles, in a population of clinical supervisors (CS) from 13 French departments of general practice.

DETAILED DESCRIPTION:
Continuing medical education is important but burdensome work for general practitioners. Current training tools have limitations and may lack the ability to engage some practitioners. Serious games are new pedagogical tools that use video games as engaging education tools. They have significant advantages in terms of efficiency and dissemination.

The aim of this work was to create a new serious game and to evaluate it in terms of efficiency and satisfaction, comparing it with a traditional method of continuing education: article reading.

We produced a prototype video game called Hygie on the 5 most common reasons of consultation in general practice using 9 articles from independent journals based on evidence (reviews by Prescrire and Minerva). We then carried out a randomized trial comparing the learning provided by a week of access to the game versus source articles, in a population of clinical supervisors (CS) from 14 French departments of general practice.

ELIGIBILITY:
Inclusion Criteria:

* to be a french general practice clinical supervisor

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3398 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Knowledge test | completed 3 to 5 weeks after the end of the intervention, i.e. 4 to 6 weeks after randomization
  Mean score at a final knowledge test
Delta knowledge | pretest before randomization, posttest 3 to 5 weeks after the end of the intervention (i.e. 4 to 6 weeks after randomization)
  Mean difference score between knowledge pretest and final knowledge test (posttest

SECONDARY OUTCOMES:
Satisfaction | one week after randomization (end of access to support)
  Satisfaction survey completed at the end of the intervention access week
Playing time | during the first week of access to support of intervention
  Time spended playing by subjects assigned to Hygie
Use in practice | completed 3 to 5 weeks after the end of the intervention, i.e. 4 to 6 weeks after randomization
  completed 3 to 5 weeks after the end of the intervention, participants answer the question "In the course of your practice, did you use the knowledge you learned through the teaching material?"

CONTACTS AND LOCATIONS:
Locations (1):
- Paris Diderot University, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: if asked
Access Criteria: requests will be considered individually

REFERENCES:
- [Derived] Jaunay LB, Zerr P, Peguin L, Renouard L, Ivanoff AS, Picard H, Griffith J, Chassany O, Duracinsky M. Development and Evaluation of a New Serious Game for Continuing Medical Education of General Practitioners (Hygie): Double-Blinded Randomized Controlled Trial. J Med Internet Res. 2019 Nov 20;21(11):e12669. doi: 10.2196/12669. PMID 31746775